CLINICAL TRIAL: NCT04984538
Title: Implementation of a Pharmacist-led Pharmacogenomic Clinical Service
Status: Withdrawn | Type: Observational
Why Stopped: Personnel Changes
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: PGX-INITIATIVE-TRHC-2020-002
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Adverse Drug Event; Drug Drug Interaction; Pharmacogenomics; Elderly
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pharmacogenomic Testing — Cheek swab as a part of routine care

SUMMARY:
Tabula Rasa HealthCare (TRHC), doing business as CareKinesis, is the first national pharmacy that provides science-based medication risk identification and mitigation technologies and services. CareKinesis utilizes medication decision support tools and pharmacists certified in geriatrics to provide pharmacy services for various healthcare organizations including PACE organizations (described above). Presently, CareKinesis services more than 35 PACE organizations, including approximately 100 PACE sites, across the United States. As a national PACE pharmacy provider since 2011, CareKinesis focuses on improving medication regimens to reduce medication-related risks while enhancing economic, clinical and humanistic outcomes. Pharmacist-led PGx clinical services and medication safety reviews are currently being offered to PACE organizations under the direction of licensed healthcare prescribers by TRHC (CareKinesis). Our aim is to extend and meticulously study PGx testing for more PACE patients and conduct a prospective preemptive PGx study to determine feasibility of implementation and effect on outcomes. After mutual agreement, these services may also be extended to other organizations where TRHC provides pharmacy services, and data will be collected with patient consent.

DETAILED DESCRIPTION:
This project aims to include patients enrolled in PACE organizations or other healthcare organizations serviced by TRHC. PGx testing will be performed by a vendor contracted by TRHC (CLIA certified). Genetic testing for CYP450 isoforms like CYP2B6, CYP2C9, CYP2C19, CYP2D6, and CYP3A5, and transporters like SLCO1B1, ABCB1, and ABCG2 will be conducted, along with other genes in individual vendors' testing panel. The results will be integrated into TRHC's proprietary CDSS (Medication Risk Mitigation Matrix, Tabula Rasa Healthcare, Moorestown, NJ). Phenotypes related to CYP450 isoforms will be used to guide pharmacists to identify drug-drug interactions (DDIs), drug-gene interactions (DGIs), and drug-drug-gene interactions (DDGIs).(16) Clinical pharmacists will translate PGx results combined with a comprehensive DDI review into actionable clinical recommendations. Prescribers will review the pharmacist's recommendation, and based on their clinical assessment will decide whether or not to implement the therapy recommendation. Endpoints like number and type of pharmacist recommendations and uptake by physicians, follow-up drug regimens, and outcomes will be collected for up to 12 months [baseline (data from the previous year), 3, 6 and 12 months post-PGx intervention] for each patient to get a longitudinal perspective of implementing PGx into CDSS systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all the following criteria will be included:

  1. Patient is enrolled in a healthcare organization where TRHC provides pharmacy services during the implementation period;
  2. Patient is able to understand, and provide informed consent to participate.

Exclusion Criteria:

* Patients with one of the following criteria will be excluded:

  1. Have taken an investigational product in the last 30 days;
  2. Current use of illicit substances;
  3. Any other medical, cognitive or physical abnormality, disease, or disorder that would prohibit the patient from completing study procedures in the judgement of the investigator and/or the prescriber.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tabula Rasa Healthcare (TRHC) partners with Programs of All-inclusive Care for the Elderly (PACE) that provides comprehensive medical and supportive services for community-dwelling persons, mostly older adults (>55 years), as an alternative to institutionalization. The aim of PACE is to improve overall quality of life in four domains (physical, psychological, social, and spiritual) using a multidisciplinary approach.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
To measure success of implementation of the PGx consultation process, including TRHC's CDSS (providing patient-specific PGx and phenotypic reviews) | 1 year
  Quantitative
Assess uptake of recommendations based on PGx is associated with improved outcomes in patients | 1 year
  Quantitative

SECONDARY OUTCOMES:
To determine usability of implementation of PGx consult during the process of medication review as measured by clinician response to survey. | 1 year
  Qualitative / Quantitative
To determine the acceptability of recommendations provided on the basis of PGx information as measured by acceptance of the recommendation and changes in prescription made after information provided. | 1 year
  Quantitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, PhD, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No